CLINICAL TRIAL: NCT03970382
Title: A Phase 1a/1b, Open-label First-in-human Study of the Safety, Tolerability and Feasibility of Gene-edited Autologous NeoTCR-T Cells (NeoTCR-P1) Administered as a Single Agent or in Combination With Anti-PD-1 to Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of Gene Edited Autologous Neoantigen Targeted TCR T Cells With or Without Anti-PD-1 in Patients With Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: PACT Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PACT-0101
Record Dates: First submitted 2019-05-06; First posted 2019-05-31 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Solid Tumor
Keywords: melanoma; HR+ breast cancer; ovarian cancer; prostate cancer; colorectal cancer; urothelial carcinoma; adoptive cell therapy; neoantigen; T cell receptor; T lymphocyte; TCR-engineered T cells; personalized cell therapy; cell therapy; immunotherapy; gene therapy; PD-1; non-small cell lung cancer; head and neck squamous carcinoma; HER2 negative breast cancer; triple negative breast cancer; IL-2
MeSH Terms: conditions — Melanoma; Ovarian Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Carcinoma, Transitional Cell; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms | interventions — Nivolumab; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NeoTCR-P1 (Experimental): Single dose of NeoTCR-P1
  Interventions: Biological: NeoTCR-P1 adoptive cell therapy
- NeoTCR-P1 plus nivolumab (Experimental): Single dose of NeoTCR-P1 plus nivolumab 480mg IV every four weeks for up to 6 doses.
  Interventions: Biological: NeoTCR-P1 adoptive cell therapy; Biological: nivolumab
- NeoTCR-P1 plus IL-2 (Experimental): Single dose of NeoTCR-P1 plus IL-2 500,000 IU/m2 SC twice daily (BID) for 7 days.
  Interventions: Biological: NeoTCR-P1 adoptive cell therapy; Biological: IL-2

INTERVENTIONS:
Biological: NeoTCR-P1 adoptive cell therapy — The investigational agent in this protocol is NeoTCR P1, an autologous adoptive T cell therapy (ACT) for patients with solid cancer. NeoTCR P1 is composed of apheresis derived CD8 and CD4 T cells that are precision genome engineered to express one autologous TCR of native sequence that targets a neoepitope (neoE) presented by human leukocyte antigen (HLA) receptors exclusively on the surface of that patient's tumor cells and not on other cells in the body.
Biological: nivolumab — Nivolumab is a human IgG4 anti-PD-1 monoclonal antibody
  Other Names: Opdivo
  Arms: NeoTCR-P1 plus nivolumab
Biological: IL-2 — IL-2 is a biologic response modifier. It is a type of protein called a cytokine.
  Other Names: Proleukin; aldesleukin; interleukin-2
  Arms: NeoTCR-P1 plus IL-2

SUMMARY:
This is a first in human, single arm, open label, Phase 1a/1b study to determine the safety, feasibility, and efficacy of a single dose of NeoTCR-P1 T cells in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented incurable or metastatic solid tumors of the following types: melanoma, UC, ovarian cancer, colorectal cancer, breast cancer (HR+), or prostate cancer.
* Disease has progressed after at least one available standard therapy or no additional curative therapies are available.
* Measurable disease per RECIST v1.1
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1
* Adequate hematologic and end organ function determined within 30 days prior to enrollment.
* Disease-specific criteria related to the specific tumor type are required.

Note: There are additional inclusion criteria. The study center will determine if you meet all of the criteria.

Exclusion Criteria:

* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, and/or inherited liver disease
* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases
* Uncontrolled or symptomatic hypercalcemia
* Pregnancy, lactation, or breastfeeding
* Prior allogeneic stem cell transplant or solid organ transplant
* Prior chimeric antigen receptor therapy or other genetically modified T cell therapy
* Active HIV, Hepatitis B, or Hepatitis C infection
* Active tuberculosis
* Severe infection within 2 weeks prior to enrollment
* Major surgical procedure within 4 weeks prior to enrollment or anticipation of need for a major surgical procedure during the study.

Note: There are additional exclusion criteria. The study center will determine if you meet all of the criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2022-08-12 (Estimated); Study Completion 2022-08-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events as defined as DLTs | 28 days
  Dose limiting toxicity (DLT) is defined as protocol-defined adverse events that occur within 28 days following infusion of Neo-TCR-P1 administered as a single agent without or with IL-2, or in combination with nivolumab.
Number of participants with adverse events as a measure of safety and tolerability of NeoTCR-P1 or NeoTCR-P1 in combination with nivolumab | 2 years
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). Cytokine release syndrome (CRS) and neurotoxicity associated with NeoTCR-P1 will be graded according to ASBMT consensus grading.
Maximum Tolerated Dose (MTD) of NeoTCR-P1 | 2 years
  The MTD is defined as the highest dose with an observed incidence of DLT in no more than one out of six patients treated at a particular dose level.
Feasibility of manufacturing NeoTCR-P1 | 2 years
  Percent of screened patients that enroll on study and receive NeoTCR-P1

SECONDARY OUTCOMES:
Maximum concentration of NeoTCR-P1 (Cmax) in the peripheral blood | 2 years
Area-under-the-concentration-vs-time-curve (AUC) in the peripheral blood | 28 days
Persistence of NeoTCR-P1 in samples of peripheral blood | 2 years
Objective Response Rate (ORR) in participants with solid tumors following infusion of NeoTCR-P1 as a single agent or in combination with nivolumab | 2 years
  ORR will be defined as Complete Response (CR) or Partial Response (PR) per RECIST v1.1, as determined by the investigator
Duration of Response mediated by neoTCR-P1 administered as a single agent or in combination with nivolumab to participants with solid tumors | 2 years
  Duration of response, defined as time from the first occurrence of a documented objective response to the time of relapse or death from any cause
Progression free survival (PFS) in participants with solid tumors following infusion of NeoTCR-P1 as a single agent or in combination with nivolumab | 2 years
  PFS is defined from date of administration of NeoTCR-P1 cell infusion to the date of disease progression per the RECIST v1.1 or death as a result of any cause. Subjects who do not meet criteria for progression by the analysis data cut-off date will be censored at their last evaluable disease assessment date
Overall survival (OS) in participants with solid tumors following infusion of NeoTCR-P1 as a single agent or in combination with nivolumab | 2 years
  OS will be measured from the date of administration of NeoTCR-P1 to the date of death. Subjects who have not died by the analysis data cut-off date will be censored at their last date of contact.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Northwestern University Medical Center, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foy SP, Jacoby K, Bota DA, Hunter T, Pan Z, Stawiski E, Ma Y, Lu W, Peng S, Wang CL, Yuen B, Dalmas O, Heeringa K, Sennino B, Conroy A, Bethune MT, Mende I, White W, Kukreja M, Gunturu S, Humphrey E, Hussaini A, An D, Litterman AJ, Quach BB, Ng AHC, Lu Y, Smith C, Campbell KM, Anaya D, Skrdlant L, Huang EY, Mendoza V, Mathur J, Dengler L, Purandare B, Moot R, Yi MC, Funke R, Sibley A, Stallings-Schmitt T, Oh DY, Chmielowski B, Abedi M, Yuan Y, Sosman JA, Lee SM, Schoenfeld AJ, Baltimore D, Heath JR, Franzusoff A, Ribas A, Rao AV, Mandl SJ. Non-viral precision T cell receptor replacement for personalized cell therapy. Nature. 2023 Mar;615(7953):687-696. doi: 10.1038/s41586-022-05531-1. Epub 2022 Nov 10. PMID 36356599
- [Derived] Levy PL, Gros A. Fast track to personalized TCR T cell therapies. Cancer Cell. 2022 May 9;40(5):447-449. doi: 10.1016/j.ccell.2022.04.013. Epub 2022 May 9. PMID 35537408